CLINICAL TRIAL: NCT03967678
Title: Omega (n)-3 PUFA Enriched Beef to Improve Circulating Lipid Concentrations and CVD Risk Markers in Adults: a Randomised Controlled Study.
Brief Title: Omega (n)-3 PUFA Enriched Beef & Health Outcomes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Dunbia, Northern Ireland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 18/WS/0149
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: CVD; Cholesterol; Metabolic Disorder; Inflammation
Keywords: enriched beef; omega; poly unsaturated fatty acids (PUFA); cholesterol; grass fed
MeSH Terms: conditions — Metabolic Diseases; Inflammation | interventions — Red Meat; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Intervention Model Description: Double blind randomised controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Beef from standard supply (Placebo Comparator)
  Interventions: Dietary Supplement: Three portions per week (690g beef (raw weight)) for 5 weeks
- n-3 enriched beef from dietary supplement finished cattle (Experimental)
  Interventions: Dietary Supplement: Three portions per week (690g beef (raw weight)) for 5 weeks
- n-3 enriched beef from grass finished cattle (Active Comparator)
  Interventions: Dietary Supplement: Three portions per week (690g beef (raw weight)) for 5 weeks

INTERVENTIONS:
Dietary Supplement: Three portions per week (690g beef (raw weight)) for 5 weeks — Lunches served in Human Intervention Studies Unit

SUMMARY:
Red meat is an integral component of the habitual diet among the UK and Irish population, with adults consuming an average of 71grams/day. Although typically high in saturated fatty acids (SFA), red meat is also an important dietary source of protein and essential nutrients including iron, zinc, B vitamins and long chain n-3 polyunsaturated fatty acids (PUFA) which provide numerous benefits to human health, particularly related to cardiovascular disease (CVD) risk. N-3 and n-6 PUFA are a family of fatty acids with important roles in cardiovascular health, and it is often recommended in dietary guidelines to replace SFA with unsaturated fats, such as PUFA. Owing to the social and economic burden of CVD, increasing the proportions of these unsaturated fatty acids, in combination with a reduction in SFA within meat, could have a large impact on CVD risk at the population level, whilst retaining the beneficial nutrients and n-3 PUFA which meat provides.

In this research, a total of 90 eligible and consenting participants will be randomly allocated to consume three portions per week of n-3 enriched beef (from either dietary supplemented or grass-fed cattle) or control beef (from standard supply). This beef will be offered within a lunchtime meal and served from the Human Intervention Studies Unit at Ulster University, Coleraine for a period of 5 weeks. A fasting blood sample will be taken before and after intervention to determine the effect the n-3 enriched beef on cholesterol concentrations, lipid profile, PUFA status and inflammation. Blood pressure, stiffness of the arteries and body shape, size and composition will also be assessed, and some health and lifestyle habits will be captured using questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Free-living, apparently healthy adults
* Aged 20+ years at recruitment
* Low oily fish consumers (<2 servings/mo), or those willing to reduce their fish consumption 1 month prior to commencing the study
* Non-smokers
* Not regularly consuming plant stanols or other n-3 enriched foodstuffs

Exclusion Criteria:

* Non-free-living adults
* Adults <20 years at recruitment
* Oily fish consumers (2 servings/mo or more)
* Current smokers
* Pregnant/lactating females (or planning to become pregnant)
* Food allergy or intolerance that would prevent consumption of the study meals
* Diagnosed with a chronic medical condition (such as diabetes; CVD; autoimmune/ inflammatory disorders; cancer)
* Prescribed cholesterol or blood pressure lowering medications
* Currently taking any fish oil-containing supplement Daily consumption of plant stanols or other n-3 enriched foodstuffs

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

PRIMARY OUTCOMES:
Cholesterol levels | Change at 5 weeks from baseline
  Plasma cholesterol measured colormetrically

SECONDARY OUTCOMES:
Lipid profile | Change at 5 weeks from baseline
  Plasma lipids measured colormetrically
Polyunsaturated fatty acid profile | Change at 5 weeks from baseline
  Serum fatty acids measured by GC-MS
Pulse Wave Velocity | Change at 5 weeks from baseline
  Measured by Sphygmocor XCEL
Blood pressure | Change at 5 weeks from baseline
  Measured by electronic blood pressure monitor
Whole body composition | Change at 5 weeks from baseline
  Measured by Dual Energy X-ray Absorptiometry
Inflammation status | Change at 5 weeks from baseline
  Measured by ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Human Intervention Studies Unit, Ulster University, Coleraine, Co.Londonderry, United Kingdom

IPD SHARING:
Plan to Share IPD: No